CLINICAL TRIAL: NCT05307380
Title: Transcultural Validation of the French Version of the Functional Pain Scale "Defense and Veterans Pain Rating Scale DVPRS"
Brief Title: Transcultural Validation of the French Version of the Functional Pain Scale "Defense and Veterans Pain Rating Scale"
Acronym: VALIDE
Status: Completed | Type: Observational
Sponsor: Benno Rehberg-Klug (Other)
Collaborators: Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Benno Rehberg-Klug, consultant anesthesiologist, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: VALIDE
Record Dates: First submitted 2022-03-04; First posted 2022-04-01 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with pain: patients with acute postoperative or post-traumatic pain or chronic pain
  Interventions: Diagnostic Test: "functional pain scale"

INTERVENTIONS:
Diagnostic Test: "functional pain scale" — French translation of the Defence and Veterans Pain Rating Scale (DVPRS)

SUMMARY:
The project will validate the French translation of the "Defense and Veterans Pain Rating Scale (DVPRS)" in multiple patient types: postoperative patients, non-surgical patients with chronic pain in the context of geriatrics, palliative care, and rehabilitation

DETAILED DESCRIPTION:
The primary objective of this study is to validate the French translation of the multidimensional "Defence and Veterans Pain Rating Scale" (= functional pain scale).

The hypothesis is that the functional pain scale is a valid measurement instrument for acute and chronic pain evaluation in a wide range of patient groups: postoperative patients, hospitalized patients with non-surgical pain (medical, oncological, rehabilitative, geriatric, palliative), and ambulatory chronic pain patients.

The primary endpoint is construct validity assessed as the association (intraclass correlation coefficient) between the pain intensity noted on the functional pain scale and on the classical NRS pain scale.

In addition to the association with the NRS, construct validity will be assessed by correlation of pain intensity noted on the functional pain scale intensity with the pain intensity score of the BPI for chronic pain patients, and the item "severe pain time" of the International Pain Outcomes Questionnaire (8) for postoperative patients.

Content validity will be assessed in a subgroup of patient by the association of the values for pain intensity (0-10) on the functional pain scale and the corresponding word descriptors. A factor analysis of all items of the functional pain scale will be performed.

Internal consistency of the functional pain scale will be tested by calculating Cronbach's alpha across all items.

Criterion validity will be assessed in patients for whom mobilisation is an important therapeutic goal as the discrimation between patients who can be mobilized and those who can't because of pain, and patients who consider their pain as tolerable and those who do not.

This discrimative ability will also be compared to the classical numeric rating scale, as it is a potential advantage of the functional pain scale. For the numeric rating scale, a large overlap in pain intensity for patients who consider their pain as tolerable and those who do not has been found(9).

Sensitivity to change will be evaluated by comparing values before and after an analgesic treatment for a subgroup of patients with an initial pain intensity of at least 4/10 on the functional pain scale. However, since patients with high pain levels will not be able to fill in the questionnaire, this is only an exploratory endpoint of this study.

Patient and caregiver evaluation of ease of use will also be evaluated, as well as patient judgement of tolerable pain levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or chronic pain, either having undergone painful surgical procedures, or having a chronic pain consultation, or being hospitalized in oncology, rehabilitative, geriatric or palliative care with painful conditions
* French-speaking and able to understand the study information
* ≥18 years of age

Exclusion Criteria:

* Inability to understand the consent form and the questionnaire, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 100 postoperative patients,
  * 50 ambulatory chronic pain patients
  * 50 hospitalized patients with non-surgical pain (medical, oncological, rehabilitative, geriatric, palliative),
  In addition, the following subgroups are planned within the total of 200 patients:
  * 30 postoperative patients with a pain intensity of at least 4 will receive the functional pain scale twice, before and after an analgesic on-demand treatment.
  * 30 patients will receive a separate sheet on which they are asked to connect the numeric pain intensity values (0-10) to the word descriptors of the functional pain scale.
  * 30 patients >75 years old
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
construct validity for acute pain | immediate after inclusion
  association (intraclass correlation coefficient) between the pain intensity noted on the functional pain scale and on the classical NRS pain scale.

SECONDARY OUTCOMES:
construct validity for chronic pain | immediate after inclusion
  correlation of pain intensity noted on the functional pain scale intensity with the pain intensity score of the BPI for chronic pain patients
Criterion validity: ability to be mobilized | immediate after inclusion
  ability to be mobilized as noted by the caregiver: the patient cannot be mobilized due to pain vs. mobilisation is possible
Criterion validity : pain intensity considered as tolerable | immediate after inclusion
  pain intensity considered as tolerable by the patient on a 0 to 10 numeric scale
Sensitivity to change | immediate after inclusion
  comparison of values before and after an analgesic treatment for a subgroup of patients with an initial pain intensity of at least 4/10 on the functional pain scale
Patient and caregiver evaluation of ease of use | immediate after inclusion
  Patient and caregiver evaluation of ease of use evaluated on a Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Benno Rehberg-Klug, MD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Hôpital du Valais, Sion, Valais
  - Hôpitaux Universitaires de Genève, Geneva

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Safran SL, Follonier D, Weber E, Vayne-Bossert P, Ahrendts U, Rehberg-Klug B. Cross-cultural adaptation and psychometric validation of the French version of the Defense and Veterans Pain Rating Scale for acute and chronic pain: a prospective clinical study. Pain Med. 2024 Oct 1;25(10):630-636. doi: 10.1093/pm/pnae049. PMID 38870517